CLINICAL TRIAL: NCT00793689
Title: Comparison of the Prognostic Value of Perioperative Parathormone Measurement and Sodium Bicarbonate Infusion Test in the Evaluation of Parathyroid Function After Total Thyroidectomy
Brief Title: Perioperative Parathormone Measurement and Sodium Bicarbonate Infusion Test After Total Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: AHEPA University Hospital (Other)
Responsible Party: John G. Yovos, Prof, Aristotle University Of Thessaloniki
Other Study IDs: APC00994614
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Hypoparathyroidism
Keywords: parathyroid; thyroidectomy; hypoparathyroidism; Parathyroid function after total thyroidectomy
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- total thyroidectomy: patients undergoing total thyroidectomy

SUMMARY:
In the study will be included patients that have undergone total thyroidectomy and do not display obvious clinical or laboratory hypoparathyroidism. On the third postoperative day and before the patient's exit from the hospital, the patient will undergo an intravenous infusion test with 35ml/m2 dilution of 8.4%(w/v) sodium bicarbonate in two minutes. Three months after the operation, if the study conditions are still met, the patient will undergo an additional parathyroid hormone (PTH) measurement and sodium bicarbonate infusion test and the parathyroid function will be evaluated again.

DETAILED DESCRIPTION:
Each patient will undergo a thorough preoperative examination for the presence of abnormalities in calcium, phosphate or magnesium metabolism as a consequence of a primary or a secondary disease.

Blood samples will be taken right before the beginning of the thyroidectomy, and 20 minutes after the end, to measure the PTH levels and to evaluate the variation rate.

On the third postoperative day and before the patient's exit from the hospital, the patient will undergo an intravenous infusion test with 35ml/m2 dilution of 8.4%(w/v) sodium bicarbonate in two minutes. Blood samples will be collected from a different vein at 0, 3, 5, 10, 30 and 60 minutes after infusion to measure PTH, calcium, phosphate and magnesium.

Three months after the operation, if the study conditions are still met, the patient will undergo an additional PTH measurement and sodium bicarbonate infusion test and the parathyroid function will be evaluated again.

In addition, the test will be performed on 50 healthy volunteers, in order to assess the response to the test of normal individuals.

ELIGIBILITY:
Inclusion criteria for the patient group

1. Patient is over 18 years old
2. Patient scheduled for total thyroidectomy
3. Patient signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures

Exclusion criteria the patient group:

1. Primary hyperparathyroidism
2. Primary hypoparathyroidism
3. Diabetes mellitus
4. Chronic Renal Failure
5. Hypoalbuminemia
6. Systematic Diseases (e.g., infections, neoplasmas)
7. Thyroid or parathyroid cancer
8. Osteoporosis
9. Drugs that influence calcium metabolism (vitamin D analogues, oral calcium supplements, biphosphonates, teriparatide, thiazide diuretics)
10. Osteomalacia
11. Neck irradiation

Inclusion criteria for the control group

1. Participant is over 18 years old
2. Participant signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures

Exclusion criteria of the control group:

1. All the above mentioned, in addition to prior thyroid surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total thyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Compare the prognostic value in the evaluation of parathyroid function of perioperative PTH measurement and sodium bicarbonate infusion test after total thyroidectomy | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: John G Yovos, MD, PhD, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Warren FM, Andersen PE, Wax MK, Cohen JI. Perioperative parathyroid hormone levels in thyroid surgery: preliminary report. Laryngoscope. 2004 Apr;114(4):689-93. doi: 10.1097/00005537-200404000-00017. PMID 15064625
- [Background] Iwasaki Y, Mutsuga N, Yamamori E, Kakita A, Oiso Y, Imai T, Funahashi H, Tanaka Y, Kondo K, Nakashima N. Sodium bicarbonate infusion test: a new method for evaluating parathyroid function. Endocr J. 2003 Oct;50(5):545-51. doi: 10.1507/endocrj.50.545. PMID 14614210